CLINICAL TRIAL: NCT01489917
Title: Comparison of A-priori Versus Provisional Heparin Therapy on Radial Artery Occlusion After Transradial Coronary Angiography and Patent Hemostasis
Brief Title: A-priori Versus Provisional Heparin on Radial Artery Occlusion After Transradial Coronary Angiography and Patent Hemostasis
Acronym: PHARAOH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Olivier F. Bertrand (Other)
Collaborators: Community Medical Center, Scranton, PA (Other); Sheth Vadilal Sarabhai General Hospital (Other)
Responsible Party: Sponsor-Investigator, Olivier F. Bertrand, Project Leader Transradial Research and Education Fund, Laval University
Organization: Laval University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PHARAOH
Record Dates: First submitted 2011-12-01; First posted 2011-12-12 (Estimated); Last update posted 2012-05-08 (Estimated); Status verified 2011-12

CONDITIONS: Coronary Artery Disease
Keywords: radial artery occlusion; hemostasis; coronary intervention; radial approach
MeSH Terms: conditions — Coronary Artery Disease; Arterial Occlusive Diseases | interventions — Heparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Compression without adjustment (No Intervention): TR band (Terumo medical) applied. The TR band is then deflated gradually till pulsatile bleeding is observed under the transparent plastic inflatable chamber and then 1-2 cc of air is placed back in the TR band chamber to stop bleeding. The band is left in place for 2 hours and not adjusted further unless patient complained of symptoms or bleeding occurred.
- Patent hemostasis & heparin (Experimental): TR-band is placed and positioned similarly to the other study arm. However, in theses cases, patency is evaluated at the time of application of the TR-band, and monitored every 15 minutes afterwards till the band is removed and hemostasis completed. After TR-band placement, if maintenance of radial artery patency is obtained, no heparin is administered and TR band is left in place for 1-hour. If radial artery patency is not maintained, a bolus of heparin 50 U/kg or a maximum of 5000 units is administered and the band is left in place for 2 hours.
  Interventions: Other: Patent hemostasis and heparin

INTERVENTIONS:
Other: Patent hemostasis and heparin — Radial artery patency is verified. If not maintained, then a bolus of heparin 50 U/kg or a maximum of 5000 units is administered and the compression (TR band) is left in place for 2 hours.
  Arms: Patent hemostasis & heparin

SUMMARY:
The Provisional Heparin TherApy on Radial Artery Occlusion after transradial coronary angiography and patent Hemostasis (PHARAOH) study compares the strategy of standard a-priori heparin use in patients undergoing transradial coronary angiography to a strategy of provisional heparin administration only if patent hemostasis is not achievable.

DETAILED DESCRIPTION:
Transradial access use for coronary angiography and intervention is increasing. Its efficacy in lowering access site complications, as well as increased patient comfort, has been proven unequivocally. One of the complications of transradial access is radial artery occlusion (RAO) that occurs with a variable incidence. It is population specific, with a higher prevalence in subsets, such as women, and patient's with small radial arteries. RAO is also known to be higher at hospital discharge and radial recanalization may spontaneously occur at later times. It is usually asymptomatic. Its main adverse impact is by limiting future transradial access from that radial artery. Since most of the patient's with atherosclerotic vascular disease may undergo several invasive procedures during their lifetime, prevention of RAO is of paramount importance.

Heparinization, during the procedure, has been shown to be of benefit in lowering the incidence of RAO. Maintaining patency of the radial artery during hemostasis, has also been shown to be effective in prevention of RAO following transradial access. As maintenance of flow has potent antithrombotic effect, it is unclear whether systemic anticoagulation is still required in all cases.

In some cases, it would be preferable to avoid heparin administration prior to coronary angiography. It is currently unknown whether it would be safe to refrain from heparin administration in case of transradial catheterization and patent hemostasis technique.

ELIGIBILITY:
Inclusion Criteria:

* all diagnostic cardiac cath patients

Exclusion Criteria:

* warfarin therapy
* previous ipsilateral TRA
* lack of consent
* abnormal (type D) Barbeau test
* scleroderma
* thrombocytopenia
* or other contraindications to heparin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 428 (Actual)
Dates: Start 2009-05; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Radial artery occlusion | At 30 days after the cathlab procedure
  Plethysmography, confirmed with duplex Doppler ultrasonography

SECONDARY OUTCOMES:
Radial artery occlusion | At 24 hours after the cathlab procedure
  Plethysmography, confirmed with duplex Doppler ultrasonography

CONTACTS AND LOCATIONS:
Overall Officials: Samir B. Pancholy, MD, Principal Investigator — TCMC, Scranton (PA, USA)
Locations (3):
- Commonwealth Medical College,, Scranton, Pennsylvania, United States
- IUCPQ, Québec, Quebec, Canada
- Sheth VS General Hospital,, Ahmedabad, India